CLINICAL TRIAL: NCT02024919
Title: Short Term Effect of Diltiazem on Myocardial Perfusion in Patients With Isolated Coronary Artery Ectasia- a Prospective Clinical Study
Brief Title: Effect of Diltiazem on Coronary Artery Ectasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Özgür Ulaş Özcan, Dr, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AnkaraU1
Record Dates: First submitted 2013-12-29; First posted 2013-12-31 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Ectasia
MeSH Terms: conditions — Coronary Aneurysm | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Diltiazem (Active Comparator): intracoronary diltiazem 5 milligrams which is diluted with 5 mL of saline
  Interventions: Drug: intracoronary administration of diltiazem
- Saline (Placebo Comparator): intracoronary saline 5 mL
  Interventions: Drug: intracoronary injection of 5 mL saline

INTERVENTIONS:
Drug: intracoronary administration of diltiazem
  Arms: Diltiazem
Drug: intracoronary injection of 5 mL saline
  Arms: Saline

SUMMARY:
Coronary artery ectasia (CAE) has been defined as localized or diffuse dilatation of epicardial coronary arteries more than 1.5 fold of adjacent normal segments. Isolated CAE constitutes minor portion of the total CAE cases, with an incidence of 0.1% to 0.79% in which coronary artery stenosis or severe valvular heart diseases are not present. CAE represents not only an anatomical variant but also a clinical constellation of coronary artery disease (CAD) like association with myocardial ischemia and acute coronary syndromes. Patients with CAE without significant coronary narrowing may still present with angina pectoris, positive stress tests, or acute coronary syndromes. Impaired epicardial and microvascular perfusion were demonstrated in ectatic coronary arteries.

Myocardial blush grading (MBG) technique has been utilized in various conditions such as acute myocardial infarction, coronary artery ectasia, syndrome X and idiopathic dilated cardiomyopathy to evaluate myocardial perfusion.

There is still no consensus for management of CAE. Previously improvement of coronary flow has been demonstrated by mibefradil in patients with slow coronary flow. A new trial is needed to explore the effect of calcium channel blockers (CCB) in isolated CAE. Diltiazem improves myocardial perfusion by blocking calcium channels in coronary arteries. This agent has been widely used in coronary catheter labs to prevent and treat no-reflow.

The current study with prospective design was therefore set up to assess whether epicardial flow and tissue level perfusion would be improved by diltiazem in myocardial regions subtended by the ectatic coronary arteries among patients with isolated CAE.

ELIGIBILITY:
Inclusion Criteria: Patients with isolated coronary artery ectasia at least 1 major epicardial coronary artery

Exclusion Criteria:

Patients with known allergy to diltiazem acute coronary syndrome left ventricular systolic dysfunction significant valvular heart disease heart failure systolic blood pressure <90 mmHg heart rate <60 atrioventricular block (grade > I) severe liver or kidney failure significant coronary artery stenosis and patients on treatment with calcium channel blockers were excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Myocardial blush grade | within 3 minutes after intracoronary diltiazem administration
  Myocardial blush grade which is a measure of myocardial perfusion will be analysed just after administration of intracoronary diltiazem.
TIMI (Thrombolysis in myocardial infarction) flow grade | Within 3 minutes after intracoronary administration of diltiazem
  TIMI (Thrombolysis in myocardial infarction) flow grade which is a measure of epicardial flow rate will be measured just after administration of intracoronary diltiazem
TIMI (Thrombolysis in myocardial infarction) frame count | within 3 minutes after intracoronary administration of diltiazem
  TIMI (Thrombolysis in myocardial infarction) frame count which is a measure of epicardial flow rate will be analysed just after administration of intracoronary diltiazem

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School Of Medicine, Department of Cardiology, Ankara, Turkey (Türkiye)